CLINICAL TRIAL: NCT03240068
Title: Protective Effects of Angiotensin-(1-7) in Peripheral Arterial Disease
Brief Title: Angiotensin-(1-7) in Peripheral Arterial Disease
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study funding ended prior to completion.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Amy Arnold, Associate Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6189
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Arterial Disease
Keywords: Renin-Angiotensin System; Inflammation; Cardiovascular; Atherosclerosis
MeSH Terms: conditions — Peripheral Arterial Disease; Inflammation; Atherosclerosis | interventions — angiotensin I (1-7); Acetates; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Angiotensin-(1-7) (Experimental): Subjects will receive intravenous infusion of five ascending doses of angiotensin-(1-7). The doses are: 1, 2, 4, 8, and 12 ng/kg/min. Each dose will be maintained for 10 minutes, for a total infusion period of 50 minutes.
  Interventions: Drug: Angiotensin 1-7
- Saline (Placebo Comparator): Subjects will receive intravenous infusion of saline that is matched in volume to the angiotensin-(1-7) arm. Saline infusion will be maintained for a total infusion period of 50 minutes.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Angiotensin 1-7 — This is a biologically active hormone of the renin-angiotensin system. It may play a beneficial role in regulation of blood pressure by dilating blood vessels and reducing inflammation.
  Other Names: Angiotensin I (1-7); Angiotensin I/II (1-7) Acetate
  Arms: Angiotensin-(1-7)
Drug: Saline — Normal saline will be used as the placebo comparator.
  Other Names: normal saline; 0.9% sodium chloride
  Arms: Saline

SUMMARY:
Peripheral arterial disease (PAD) affects over 8 million individuals in the United States alone. This is a form of atherosclerosis in which plaques preferentially build up inside the arteries of the legs to limit blood flow. These patients are at high risk for heart attack and stroke, with at least half dying from coronary artery disease. Our understanding of the causes of PAD remains incomplete. The renin-angiotensin hormone system is one mechanism known to contribute to atherosclerosis. Pharmacologic blockade of the hormone angiotensin II is beneficial in forms of atherosclerosis, including peripheral arterial disease, to improve blood vessel damage and functional outcomes. These therapies also increase circulating levels of angiotensin-(1-7), a hormone that dilates blood vessels. Angiotensin-(1-7) improves blood vessel function and reduces inflammation to protect against atherosclerosis in animal models; however, there are no clinical data in patients with atherosclerosis. The overall goal of this project is to examine the cardiovascular effects of angiotensin-(1-7) in PAD.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled, crossover study to determine if acute intravenous Ang-(1-7) infusion can reduce systemic inflammation and improve measures of leg blood flow in subjects with PAD. The investigators will also measure for changes in blood pressure and circulating hormones in response to angiotensin-(1-7) infusion. This is an outpatient study that will be conducted in the Clinical Research Center at the Penn State Milton S. Hershey Medical Center.

Subjects with PAD will participate in a screening visit, and if eligible, in two separate study visits in which they will receive intravenous angiotensin-(1-7) or saline infusion. Each study visit will last approximately 4 hours, with at least one week of washout between study visits. During study visits, subjects will be instrumented with two intravenous catheters (one for drug infusion and one for blood sampling), arm and finger blood pressure cuffs, sticky patches to measure heart rate, a belt around the stomach to measure breathing, an ultrasound probe on each leg to measure blood flow, a probe on the ear to measure blood oxygen saturation, a probe on each calf muscle to measure oxygen levels, and probes on the skin to measure temperature and blood flow. The investigators will obtain baseline measures of blood pressure and heart rate and collect blood samples to measure hormones in the blood. After baseline measurements, the investigators will infuse angiotensin-(1-7) or saline for 50 minutes. Finger cuff blood pressure, leg blood flow, and calf muscle oxygen levels will be measured continuously during infusions. The investigators will measure blood pressure and heart rate and collect blood samples at the end of the infusion period.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or Female
* Age: 21-80 years of age
* Diagnosed with PAD (e.g. ankle-brachial index below 0.9)
* Fontaine stage II or less (no rest pain)
* Capable of giving informed consent
* Fluent in written and spoken English

Exclusion Criteria:

* Age less than or equal to 20 years or greater than or equal to 81 years
* Pregnant or nursing woman
* Decisional impairment
* Prisoners
* Alcohol or drug abuse
* Evidence of type I or type II diabetes (fasting glucose >126 mg/dl or use of anti-diabetic medications)
* History of serious cardiovascular disease (e.g. myocardial infarction within 6 months, symptomatic coronary artery disease, presence of angina pectoris, significant arrhythmia, congestive heart failure, deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis, hypertrophic cardiomyopathy) or cerebrovascular disease (e.g. cerebral hemorrhage, stroke, transient ischemic attack).
* History or presence of immunological or hematological disease
* Impaired hepatic function [aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels > 2 times the upper limit of normal range)
* Impaired renal function (serum creatinine >2.0 mg/dl)
* Anemia
* Treatment with serotonin-norepinephrine reuptake inhibitors (SNRI) or norepinephrine transporter (NET) inhibitors
* Treatment with phosphodiesterase-5 inhibitors
* Treatment with anticoagulants
* Treatment with chronic systemic glucocorticoid therapy (>7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1-month preceding the study
* Inability to give, or withdraw, informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Leg Blood Flow | 50 minutes
  The change in measures of leg blood flow (e.g. femoral blood flow and conductance, calf muscle oxygen saturation) following angiotensin-(1-7) versus saline infusion.
Inflammatory Markers | 50 minutes
  The change in blood levels of inflammatory markers C-Reactive Protein and Interleukin-6 following angiotensin-(1-7) versus saline infusion.

SECONDARY OUTCOMES:
Blood Pressure | 50 minutes
  The change in arm and finger cuff blood pressure following angiotensin-(1-7) versus saline infusion.
Heart Rate | 50 minutes
  The change in heart rate following angiotensin-(1-7) versus saline infusion.

OTHER OUTCOMES:
Renin-Angiotensin System Hormones | 50 minutes
  The change in circulating levels of renin-angiotensin system hormones (e.g. plasma renin activity, angiotensin peptides, aldosterone) following angiotensin-(1-7) versus saline infusion.
Nitric Oxide Bioavailability | 50 minutes
  The change in circulating levels of nitrate and nitrite following angiotensin-(1-7) versus saline infusion.
Lipids | 50 minutes
  The change in circulating lipids (e.g. cholesterol, triglycerides) following angiotensin-(1-7) versus saline infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Arnold, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No